CLINICAL TRIAL: NCT05649007
Title: Post-marketing Surveillance Study of the Saphir Stem in Primary Hip Surgery
Status: Recruiting | Type: Observational
Sponsor: Gruppo Bioimpianti S.r.l. (Industry)
Responsible Party: Sponsor
Other Study IDs: PRCS202201
Record Dates: First submitted 2022-12-02; First posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Arthropathy of Hip
MeSH Terms: interventions — Prostheses and Implants

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: hip arthroplasty with prosthesis — Use of femoral stem and acetabular cup for hip arthroplasty

SUMMARY:
Post-market clinical follow up investigation on the use of saphir stem and FIN Cup or Dualis system in the treatment of pathologies requiring hip arthroplasty. The main object of the clinical investigation is the evaluation of long term survival rate of Saphir stem.

DETAILED DESCRIPTION:
The main object of the clinical investigation is the evaluation of Stem (SAPHIR) survival rate. The post market clinical follow up will also consider as further seconday endpoints: improvement of paient function, quality of life, safety of device (intended as possible adverse events related to the use of the prosthesis)

ELIGIBILITY:
Inclusion Criteria:

* patients>18 years
* Candidate for primary total hip replacement with femoral stem and acetabular cup
* if ostheoarthritis patients aged 18 to 85 years
* if femoral neck fracture patients aged 18 to 90 years
* patients with social security scheme
* patients understands the condition of the study and is willing to partecipate for the duration of the clinical investigation
* patients who gavee consent to partecipare in the clinical investigation

Exclusion Criteria:

* <18 years
* if female, pregnant
* patient who has already had primary hip surgery on the same side
* local or disseminated neoplastic disease
* inability to understand the study and agree to partecipate
* patients cancelling partecipation before surgery
* patients under guardianship or curatorship
* patients without a social security scheme
* patients refusing to partecipate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: please see inclusion/exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 630 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2035-09-30 (Estimated); Study Completion 2036-09-30 (Estimated)

PRIMARY OUTCOMES:
stem survival rate | 1 year, 3 years, 5 and 10 years
  Kaplan Meier survival analysis

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Giordano, medicine, Principal Investigator — Hopital Ducuing
Locations (1):
- Hopital Ducuing, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided